CLINICAL TRIAL: NCT03326414
Title: Influence of Different PEEP Levels and Different Tidal Volumes on Regional Pulmonary Function in Patients Undergoing Robot Assisted Prostatectomy Detected by Electrical Impedance Tomography
Brief Title: Influence of Different PEEP Levels and Tidal Volumes on Regional Lung Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANA-UKE-PV5538
Record Dates: First submitted 2017-08-28; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Ventilation; Newborn, Abnormal
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Intervention Model Description: 40 patients are to be investigated during the project. In phase one 20 patients are ventilated with constant PEEP of 10mbar and the tidal volume is set to 4-5ml/kg IBW or 8-10ml/kg IBW respectively. In phase two further 20 patients are ventilated with a constant tidal volume of 8ml/kg IBW and the PEEP is set to 3mbar or 12mbar respectively.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Constant PEEP - low tidal volume (Other): PEEP is 10mbar, tidal volume is set to 4-5ml/kg IBW
  Interventions: Procedure: Constant PEEP - low tidal volume
- Constant PEEP - high tidal volume (Other): PEEP is 10mbar, tidal volume is set to 8-10ml/kg IBW
  Interventions: Procedure: Constant PEEP - high tidal volume
- constant tidal volume - low PEEP (Other): tidal volume is 8ml/kg IBW, PEEP is set to 3mbar
  Interventions: Procedure: constant tidal volume - low PEEP
- constant tidal volume - high PEEP (Other): tidal volume is 8ml/kg IBW, PEEP is set to 12mbar
  Interventions: Procedure: constant tidal volume - high PEEP

INTERVENTIONS:
Procedure: Constant PEEP - low tidal volume — The respirator is set according to study protocol
  Arms: Constant PEEP - low tidal volume
Procedure: Constant PEEP - high tidal volume — The respirator is set according to study protocol
  Arms: Constant PEEP - high tidal volume
Procedure: constant tidal volume - low PEEP — The respirator is set according to study protocol
  Arms: constant tidal volume - low PEEP
Procedure: constant tidal volume - high PEEP — The respirator is set according to study protocol
  Arms: constant tidal volume - high PEEP

SUMMARY:
Mechanical ventilation is indispensable for most of surgical interventions but can induce lung injury even in pulmonary healthy patients. This can lead to postoperative pulmonary complications. These adverse effects could be prevented by a better monitoring of intraoperative lung function. Electrical impedance tomography is able to visualize aeration within the lung in real time.

The planned study investigates the influence of different levels of positive endexspiratory pressure and different tidal volumes on the aeration.

DETAILED DESCRIPTION:
Available perioperative parameters to set mechanical ventilation parameters represent only global lung function. But to reduce postoperative pulmonary complications induced by mechanical ventilation a better monitoring of intraoperative lung function seems to be crucial, that provides more regional information of lung collapse or over distention.

By application of small currents via electrodes around the thorax and measuring of the resultant resistance the electrical impedance tomography (EIT) can determine the level of aeration of the lung in a cross sectional plane. The EIT device used in this study calculates the percentage of the investigated lung area that can be defined as over distended or collapsed respectively. In these sections the change of resistance within a respiration cycle is reduced compared to well ventilated areas are therefore called silent spaces. Silent spaces located ventral are termed non-dependent (NSS) and silent spaces located dorsal are termed dependent (DSS). Based on this information the clinician is able to set the respirator in a more lung protective manor.

To better understand the influence of positive endexspiratory pressure (PEEP) and tidal volume (Vt) on reginal lung function we are going to carry out the presented study.

40 patients undergoing robot assisted prostatectomy should be enrolled in a study that consists of two phases. In the first phase 20 patients are ventilated with constant PEEP (10mbar) and in ten patients each the Vt is set to 5 or 12ml/kg ideal body weight. In the second phase in further 20 patients the Vt is set to 8ml/ kg ideal bodyweight and the PEEP is 3 or 12mbar in one half of the patients. Under the different ventilation settings the NSS and DSS, the oxygenation index and lung compliance will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* scheduled for robot assisted prostate ectomy

Exclusion Criteria:

* body mass index >35 kg/m²
* chronic obstructive lung disease (GOLD III or IV)
* obstructive sleep apnoe syndrome
* planned or unplanned admission to intensive care unit for prolonged ventilation
* mechanical ventialtion within the last 30 days
* lung operation in the past
* other lung disease that impairs activity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is carried out in patients undergoing prostatectomy
Enrollment: 40 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change of "dependent silent spaces" (DSS) and "non-dependent silent spaces" (NSS) | measurement of DSS and NSS are carried out prior to induction of anesthesia, 10 minutes after induction, 30 minutes after after installation of capnoperitoneum, 10 minutes after skin closure, 15 minutes after arrival at the PACU
  The change of silent spaces under different ventilator settings during surgery is investigated.

SECONDARY OUTCOMES:
Oxygenation index | prior to induction of anesthesia, 10 minutes after induction, 30 minutes after installation of capnoperitoneum, 10 minutes after skin closure, 15 minutes after arrival at the PACU
  The partial pressure of oxygen is determined at every point of measurement and the value is devided by inspiratory oxygen fraction
complinace of the respiratory system | 10 minutes after induction, 30 minutes after capnoperitoneum applied, 10 minutes after skin closure
  The compliance of the respiratory system (ml/mbar) is mesured by the respirator during mechanical ventilation

OTHER OUTCOMES:
postoperative pulmonary complicaitons | postoperative pulmonary complications apearing within 7 days after surgery
  postoperative complications like pneumonia, reintubation and need for non-invasive ventilation are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Reuter, MD, Study Director — Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Hospital Hamburg-Eppendorf, Germany
Locations (1):
- Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not planned to share data with other researchers except data published within an article.

REFERENCES:
- [Background] Canet J, Sabate S, Mazo V, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P; PERISCOPE group. Development and validation of a score to predict postoperative respiratory failure in a multicentre European cohort: A prospective, observational study. Eur J Anaesthesiol. 2015 Jul;32(7):458-70. doi: 10.1097/EJA.0000000000000223. PMID 26020123
- [Background] Ukere A, Marz A, Wodack KH, Trepte CJ, Haese A, Waldmann AD, Bohm SH, Reuter DA. Perioperative assessment of regional ventilation during changing body positions and ventilation conditions by electrical impedance tomography. Br J Anaesth. 2016 Aug;117(2):228-35. doi: 10.1093/bja/aew188. PMID 27440635